CLINICAL TRIAL: NCT00987363
Title: Phase II Clinical Trial of Therapeutic Angiogenesis With Mononuclear Cells Autologous Bone Marrow in Patients With Chronic Ischemia Diabetics Critical Limb (CLI) no Revascularization.
Brief Title: Intraarterial Infusion of Autologous Bone Marrow in Diabetic Patients With Chronic Ischemia of Lower Limbs (CLI) no Revascularization
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMMo/ICPD/2008; 2008-004064-39 (EudraCT Number)
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2014-11

CONDITIONS: Critical Limb Ischemia (CLI); Diabetic Foot
Keywords: critical limb ischemia (CLI); diabetic foot; bone marrow derived mononuclear cells; cell therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose (1x10 E8) (Experimental): Dose of 1x10 E8 autologous bone marrow-derived mononuclear cells
  Interventions: Other: Intraarterial infusion of autologous bone marrow cells
- Intermediate dose (5x10 E8) (Experimental): Dose of 5x10 E8 autologous bone marrow-derived mononuclear cells
  Interventions: Other: Intraarterial infusion of autologous bone marrow cells
- High dose (1x10 E9) (Experimental): Dose of 1x10 E9 autologous bone marrow-derived mononuclear cells
  Interventions: Other: Intraarterial infusion of autologous bone marrow cells
- Control (No Intervention): Conventional treatment established by the good clinical practice

INTERVENTIONS:
Other: Intraarterial infusion of autologous bone marrow cells — Autologous bone marrow-derived mononuclear cells will be infused by an intraarterial catheter into de ischemic limb. The number of infused cells will be 1x10 E8, 5x10E8 and 1x10 E9 in the low,intermediate and high dose arms respectively
  Arms: High dose (1x10 E9); Intermediate dose (5x10 E8); Low dose (1x10 E8)

SUMMARY:
The aim of the study is to evaluate the safety and feasibility of autologous bone marrow mononuclear cells autologous administered intra-arterially in the affected limb of diabetic patients with chronic critical ischemia of the lower limbs (CLI) without possibility of revascularization or other therapeutic alternatives.

The trial hypothesis we propose consists of mononuclear cells of bone marrow providing progenitor cells with regenerative capacity and secrete also several angiogenic factors, and their implantation into ischemic tissues with both elements should contribute to angiogenesis and tissue regeneration with recovery of the circulation in the affected limb

DETAILED DESCRIPTION:
Phase II Clinical Trial, a prospective, multicenter, open, randomized, parallel-group controlled with three dose levels.

The study population will consist of a total of 60 diabetic patients with chronic critical ischemia of one leg (CLI) and no possibility of revascularization. In the experimental group will include a total of 45 patients divided into three dose levels, 15 patients in each level (increasing doses of mononuclear cells of bone marrow evenly) and 15 patients in control group (no cell therapy). Patients will be randomly assigned to either the control group or to any of the three experimental groups in which the dose of mononuclear cells of bone marrowo will be:

* Group 1(15 patients): no cell therapy.
* Group 2(15 patients): 1x108 mononuclear cells of bone marrow
* Gropu 3(15 patients): 5x108 mononuclear cells of bone marrow
* Group 4(15 patients): 1x109 mononuclear cells of bone marrow The cell therapy medicinal product shall be administered in all cases intraarterially.

Patients were evaluated by clinical, radiological and angiologist methods. This is a randomized controlled trial in which the safety and feasibility of cell therapy medicinal product shall be measured by comparing the response variables after treatment compared to baseline prior to implementation. Secondarily the results obtained are compared with each of the dose groups.

Patients will receive in a concomitant way the drug treatment established by the good practice, so it would certainly be possible that some improvement occurs due to drug treatment.

The primary variable is the improvement in the vascularización of the treated limb determined by clinical, angiologic and angiographic parameters.

It is estimated that the inclusion period lasts between twelve and eighteen months with twelve months follow-up. Therefore the total study duration range between twenty-four and thirty months from the inclusion of the first patient to the end of the follow-up of the last patient included.

Objectives of the study:

- Main objective: To evaluate the safety and feasibility of mononuclear cells of autologous bone marrow administered intra-arterially in the affected limb of diabetic patients with chronic critical ischemia of the lower limbs without possibility of revascularization or other therapeutic alternatives.

Secondary objectives:

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or 2 diabetes mellitus
2. Grade II-III Rutherford-Becker peripheral vascular disease affecting at least one limb
3. Arterial obstruction(s) located at infrapopliteal level
4. No options of endoarterial or surgical revascularization
5. Life expectancy more than 2 years
6. Unlikelihood of major amputation of the leg during the next 12 months
7. Normal analytical parameters in blood: leucocytes>3000/micoL, neutrophils>1500 microL, Hb>10mg/dl, platelets>100000 microL,AST and ALT<2.5 standard value, creatinin<2.5 mg/dl
8. Written informed consent
9. Negative pregnancy test when applicable

Exclusion Criteria:

1. History of neoplasm or hematological disease
2. Uncontrolled high blood pressure (>180/110)
3. Severe cardiac insufficiency (NYHA IV) or ejection fraction<30%
4. Malignant ventricular arrythmia
5. Deep venous thrombosis during the last 3 months
6. Active bacterial infection
7. Treatment with hyperbaric oxygen, vasoactive drugs, Cox-II inhibitors or antiangiogenic agents
8. Body mass index > 40
9. Alcoholism
10. Proliferative retinopathy
11. HIV, HBV or HCV viral infection
12. Stroke or myocardial infarction during the last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 24 h, 1,3 ,6 ,9 and 12 months
AngioRNM and/or AngioTC changes | baseline and 12 months

SECONDARY OUTCOMES:
Clinically objective improvement in the ischemic limb | 1, 3, 6, 9 and 12 months
  (Ankle/brachial index, transcutaneous oxygen pressure, degree of Rutherford-Becker, greater ulcer size and perimeter calf muscle)

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Herrera, MD, PhD, Study Chair — Hospital Universitario Reina Sofia de Cordoba; Francisco Tadeo Gomez, MD, PhD, Principal Investigator — Hospital Virgen del Rocio; Jose Patricio Linares, MD, PhD, Principal Investigator — Hospital Universitario San Cecilio; Diego Martinez, MD, PhD, Principal Investigator — Hospital Universitario Morales Messeguer; Vicente García, MD,PhD, Principal Investigator — University Hospital Virgen de las Nieves; Antonio Chacon, MD, PhD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (5):
- Spain (5):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario Virgen de la Nieves, Granada
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen del Rocio, Seville